CLINICAL TRIAL: NCT01389583
Title: A Phase II Study of AUY922, a Novel HSP Inhibitor, in Patients With Advanced GIST Failed to or Intolerance of Imatinib and Sunitinib Therapy
Brief Title: A Study of AUY922 for GIST(Gastrointestinal Stromal Tumor) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Mackay Memorial Hospital (Other); Taichung Veterans General Hospital (Other); China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2211
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2013-09

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: GIST(Gastrointestinal stromal tumor); HSP(Heat Shock Protein); Biomarker
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AUY922 (Experimental): AUY922
  Interventions: Drug: AUY922

INTERVENTIONS:
Drug: AUY922 — 70 mg/m2 60-min i.v. infusion weekly

SUMMARY:
A Phase II Study of AUY922, Novel HSP Inhibitor, in Patients with Advanced GIST Failed to or Intolerance of Imatinib and Sunitinib Therapy

Primary endpoint:

•The primary endpoint of this study is to assess disease control rate (complete response + partial response + stable disease≧4 months) of AUY922 in patients with advanced GIST failed to imatinib and sunitinib

Secondary endpoints:

* To determinate the objective response rate (ORR, complete response + partial response)
* To determinate the time to tumor progression (TTP)
* To evaluate the safety and toxicity profiles of AUY922
* To evaluate the pharmacokinetics profile of AUY922 in Taiwan GIST population
* To access the pharmacodynamic effect of AUY922 on HSP client proteins in blood and tumor if feasible , i.e. HSP70, in Taiwan GIST population
* To access the tissue biomarkers pre-treatment and 4wks post treatment if feasible, i.e. HSP70, c-KIT, PDGFRA mutation, ...etc in Taiwan GIST population

Exploratory endpoints:

•PET imaging; sSUVmax

DETAILED DESCRIPTION:
This is an open-label; pharmacokinetic and pharmacodynamic phase II study of AUY922 in patients with advanced GIST failed to or intolerance of imatinib and sunitinib therapy. AUY922 is a novel HSP90 inhibitor and will be administered at dose of 70 mg/m2 i.v. infusion on D1 every week. The Simon one sample two-stage minimax design was used with 15 suitable patients to be accrued to the first stage. If at least two patients meet our primary endpoint (complete response＋partial response＋stable disease≧4 months), an additional 10 patients would be recruited to the second stage. AUY922 would be considered active in this patient population, if there were more than 5 cases of non-progressive disease in the total cohort of 25 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven CD117-positive and/or c-kit or PDGFR mutation gastrointestinal stromal tumor (GIST), which is metastatic or unresectable, locally advanced, and have failed to or intolerance of prior imatinib and sunitinib treatment
2. At least one measurable lesion according to the RECIST criteria (version 1.1)
3. Aged between 20-75 years
4. With Eastern Cooperative Oncology Group (ECOG) performance score 0-2.
5. Life expectancy ≥ 4 months
6. At least 4 weeks apart from prior systemic (including chemotherapy, approved targeted therapy or investigational agent) and surgical treatment, and recovery from all prior treatment-related toxicity to grade < 1 according to Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
7. With adequate organ and marrow function as defined below:

   * WBC ≥ 3.00 × 103/ mm3 and absolute neutrophil count ≥ 1.50 × 103/ mm3
   * Platelet count ≥ 100.0 × 103/mm3
   * Hemoglobin level ≥ 9 gm/dL
   * Serum creatinine (Cr) ≦1.5 x UNL or eGFR ≥ 60 ml/min (by Cockroft-Gault method)
   * Serum bilirubin ≤ 1.5 x UNL , ALT ≤ 2.5x UNL. If obstructive jaundice with proper drainage, serum bilirubin ≤ 3 x UNL is acceptable.
8. Women of childbearing potential and men must agree to use accepted methods of contraception during the course of the study and at least 3 months after last dose of treatment
9. Willing to have tumor biopsy at screening (all patients) and able to comply with study requirement at 4 weeks post treatment
10. With ability to understand and the willingness to sign Informed Consent Form.

Exclusion Criteria:

1. Have received imatinib or sunitinib, chemotherapy, any investigational agents or participate in any investigational drug study within 28 days before enrolment
2. Have major surgery within 28 days before enrolment (diagnostic biopsy or line placement is not considered major surgery)
3. With active multiple cancers or history of other malignancy within the last three years, except treated curable non-melanoma skin cancer, in-situ cervical cancer, Dukes' A colorectal cancer.
4. With known CNS metastasis
5. Symptoms of heart failure or greater to Class III (by NYHA criteria) or history of uncontrolled dysrrhythmias
6. Sinus bradycardia (resting heart rate <50 beats/min) secondary to intrinsic conduction system disease; Patients with sinus bradycardia secondary to pharmacologic treatment may enrol if they are allowed to withdraw the treatment and can result in normalization of the resting heart rate to within normal limits
7. Myocardial infarction or active ischemic heart within 6 months
8. Screening QTc >450 msec in males; QTc >470 msec in females, or previous history of QTc prolongation while taking other medications
9. Presence of active infection or systemic use of antimicrobials within 72 hours prior to enrolment
10. Treatment with therapeutic doses of coumadin-type anticoagulants. [Maximum daily dose of 2mg, for line patency permitted]
11. Patients who are unable to comply protocol requirement, i.e. tumor tissue sampling or blood sampling for pharmacodynamic and pharmacokinetics study
12. Patients who have know hypersensitivity or prior therapy of any HSP90 inhibitor compound or its derivatives

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2011-10; Primary Completion 2015-05 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
disaese control rate | 4 months
  The primary endpoint of this study is to assess disease control rate (complete response + partial response + stable disease≧4 months) of AUY922 in patients with advanced GIST failed to imatinib and sunitinib

SECONDARY OUTCOMES:
response rate | 3 years
  * To determinate the objective response rate (ORR, complete response + partial response)
  * To determinate the time to tumor progression (TTP)
  * To evaluate the safety and toxicity profiles of AUY922
  * To evaluate the pharmacokinetics profile of AUY922 in Taiwan GIST population
  * To access the pharmacodynamic effect of AUY922 on HSP client proteins in blood and tumor if feasible , i.e. HSP70, in Taiwan GIST population
  * To access the tissue biomarkers pre-treatment and 4wks post treatment if feasible, i.e. HSP70, c-KIT, PDGFRA mutation, ...etc in Taiwan GIST population

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, M.D.,Ph.D, Principal Investigator — National Health Research of Institutes, Taiwan Cooperative Oncology Group
Locations (1):
- National Health Research of Institutes, Taiwan Cooperative Oncology Group, Tainan, Taiwan